CLINICAL TRIAL: NCT05423886
Title: The Effectiveness of Personalized Colorectal Cancer Screening Based on Fecal Hemoglobin Concentration
Acronym: PERFECT-FIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Esther Toes-Zoutendijk (Other)
Responsible Party: Sponsor-Investigator, Esther Toes-Zoutendijk, Dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: WO 19-44
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention arm receives their screening invitation within 1,2 or 3 years, depending on their previous fecal Hemoglobin concentration. The control arm receives their screening invitation in 2 years (current practice).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants receive a personalized screening invitation interval (1,2 or 3 years) based on their fecal Hemoglobin concentration of the negative fecal immunochemical test in previous round.
  Interventions: Other: Personalized screening invitation interval
- Control arm (No Intervention): Participants receive a standard screening invitation interval (2 years).

INTERVENTIONS:
Other: Personalized screening invitation interval — Time to receive the next invitation for fecal immunochemical testing screening, will depend based on individuals risk determined by fecal Hemoglobin concentration
  Arms: Intervention arm

SUMMARY:
We aim to improve the yield and effectiveness of the Dutch colorectal cancer screening program by using a personalized screening strategy based on fecal Hemoglobin concentration in previous screening round for participants with a negative fecal immunochemical test (FIT).

DETAILED DESCRIPTION:
A fecal Hemoglobin concentration just below the cut-off of the fecal immunochemical test (FIT) is associated with a higher risk for the detection of colorectal cancer of advanced adenomas at consecutive screenings. Individuals with these higher fecal Hemoglobin concentrations may benefit from shorter screenings interval, whereas individuals without any fecal Hemoglobin concentrations could benefit from longer screening intervals.

A randomized controlled trial will be conducted within the national CRC screening program among individuals with a negative FIT in the previous screening round. Individuals in the intervention arm will receive an invitation after 1, 2, or 3 years depending on their fecal Hemoglobin concentration in the previous round, whereas individuals in the control arm will receive an invitation after 2 years according to current practice.

The overall aim of this study is to improve the balance between harms and benefits of CRC screening, by using a personalized approach based on fecal Hemoglobin concentration at previous screening. More specifically, this study has three goals:

1. Evaluate the superiority of risk-based FIT screening in a randomized controlled study embedded in a running national screening program;
2. Evaluate the feasibility and acceptability of risk-based FIT screening in a national screening program;
3. Estimate the long-term effect of personalized screening versus uniform screening.

To achieve these goals a randomized controlled trial, focus groups and microsimulation modelling will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Previous negative FIT (below the cut-off of 47 microgram per gram feces)

Exclusion Criteria:

* Previously tested with FIT cut-off of 15 microgram per gram feces

Ages: 56 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Detection rate of colorectal cancer and advanced adenomas | 6 months after the last invitation
  Number of colorectal cancers and advanced adenomas per screened individual

SECONDARY OUTCOMES:
Acceptability | 6 months after the last invitation
  Number of individuals participating in personalized FIT screening

CONTACTS AND LOCATIONS:
Overall Officials: Iris Lansdorp-Vogelaar, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Outcomes of the study will be stored in the national screening information system, owned by a third-party sources. Data cannot be publicly shared.

REFERENCES:
- [Derived] Breekveldt ECH, Toes-Zoutendijk E, de Jonge L, Spaander MCW, Dekker E, van Kemenade FJ, van Vuuren AJ, Ramakers CRB, Nagtegaal ID, van Leerdam ME, Lansdorp-Vogelaar I. Personalized colorectal cancer screening: study protocol of a mixed-methods study on the effectiveness of tailored intervals based on prior f-Hb concentration in a fit-based colorectal cancer screening program (PERFECT-FIT). BMC Gastroenterol. 2023 Feb 22;23(1):45. doi: 10.1186/s12876-023-02670-1. PMID 36814185